CLINICAL TRIAL: NCT00916890
Title: Chronic Administration of Opioids in Cancer Chronic Pain:an Open Prospective Study on Efficacy, Safety and Pharmacogenetic Factors Influence.
Brief Title: Prospective Study About Clinical and Pharmacogenetic Safety of Opioid Use for Chronic Pain
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulties in patients enrolment
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-SM-1-Op-Cancer
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Pain
Keywords: Opioid pharmacogenetics; Opioid pharmacokinetic; Long-term opioid treatment; Cancer pain
MeSH Terms: conditions — Chronic Pain; Cancer Pain | interventions — Morphine; Oxycodone; Fentanyl; Buprenorphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral extended-release morphine (Active Comparator)
  Interventions: Drug: Morphine
- Oral extended-release oxycodone (Active Comparator)
  Interventions: Drug: Oxycodone
- Transdermal fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl
- Transdermal buprenorphine (Active Comparator)
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Morphine — After a titration phase with fast-release oral morphine, once the optimal dosage (no side effects and less than two rescue doses per day) is reached, an equipotent dose of oral sustained-release morphine will be randomly assigned to a patient.
  Arms: Oral extended-release morphine
Drug: Oxycodone — After a titration phase with fast-release oral morphine, once the optimal dosage (no side effects and less than two rescue doses per day) is reached, an equipotent dose of oral extended-release oxycodone will be randomly assigned to a patient.
  Arms: Oral extended-release oxycodone
Drug: Fentanyl — After a titration phase with fast-release oral morphine, once the optimal dosage (no side effects and less than two rescue doses per day) is reached, an equipotent dosage of transdermal fentanyl will be randomly assigned to a patient.
  Arms: Transdermal fentanyl
Drug: Buprenorphine — After a titration phase with fast-release oral morphine, once the optimal dosage (no side effects and less than two rescue doses per day) is reached, an equipotent dosage of transdermal buprenorphine will be randomly assigned to a patient.
  Arms: Transdermal buprenorphine

SUMMARY:
Aim of this project is to customize the choice of the strong opioid in the treatment of cancer chronic pain through the identification of patient clinical history and pain characteristics, moreover in the analysis the investigators will also correlate the clinical efficacy and safety of opioid treatment with pharmacokinetic and pharmacogenetic patterns in order to identify variables able to predict the efficacy of the treatment or the patient susceptibility towards a specific treatment.

Furthermore with this study the investigators want to identify the pharmacogenomic characterization responsible for pharmacokinetic variability in the conversion between morphine and other opioids, in order to validate the currently available conversion tables from a pharmacokinetic viewpoint, estimating the influence of the most common genetic polymorphisms, and if this characterization could be useful and cost-effective. This study will also focus on the specific clinical-pharmacological response in the elderly and between male and female and on the interactions between opioids and those anticonvulsant and antidepressant drugs routinely used in the pain therapy (study of pharmacovigilance).

DETAILED DESCRIPTION:
Pain continues to be a major problem in patients with cancer, affecting 25% to 30% of patients with recently diagnosed cancers. The incidence of pain in advanced stages of cancer approaches 70% to 80%. There are a number of reasons that patients with cancer experience chronic pain either related to the disease itself or to its treatment.

Cancer can spread by metastasis or direct invasion, and 90% of patients with metastasis to osseous structures report pain. Patients with cancer can have neuropathic pain due to direct compression of nerves or plexus or spinal cord involvement.

Inadequate treatment and undertreatment are associated with increased pain scores, decreased functional ability, and increased depression and anxiety.

Opioid administration though proven to be effective still meets with resistance from both healthcare operators, who are seldom willing to prescribe these drugs, and patients, who tend to not take them because of many false beliefs still related to opioids.

It is well demonstrated by the literature that opioids are effective in controlling both acute and chronic pain of nociceptive and/or neuropathic origin. Switching type of opioid and/or administration routes (e.g., from oral to neuraxial) is also known to be an important factor in long-term treatment: appropriate conversion tables elucidating drug equipotence and different potency in base of administration route for the different opioids currently available have therefore been devised and validated in the clinical setting.

There have been several attempts to define guidelines for treatment protocols and even recent meta-analyses indicate that morphine should remain the gold standard. However, a general consensus is still lacking, as opioid management depends not only on the type and cause of pain, but also on the patient's history, the pain characteristics and genetic patterns. Which, if any, is the best opioid, in relation with previous characters, to start systemic treatment remains therefore debated. The different effects that different opioids have on spinal cord sensitization as a result of continuous peripheral nociceptive stimulus in long term administration have also been partially investigated.

Current pharmacogenetic publications analyze the pharmacokinetic behavior of opioids in short-term administration, but studies are still lacking on how the pharmacokinetics and analgesic effect vary after repeated administrations of opioids, especially through direct comparison with clinical response. Genetic studies showed differences in the results of opioid treatment related to the variability of the genes that have a role in the pharmacodynamic and pharmacokinetics of opioids. Regardless these studies, the literature has not yet investigated how quantitative and qualitative variability of gene products can influence the efficacy or the toxicity of a specific opioid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult oncologic patients (>= 18 years old)
* Chronic peripheral neuropathic and/or nociceptive pain
* Written informed consent

Exclusion Criteria:

* Pediatric patients
* Mental impaired patients
* Substance abuse disorder
* Opioid allergy
* History of opioids use or addiction
* Severe immunodeficiency, severe renal impairment, severe liver disease
* Cachectic state
* HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2009-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To identify the drug with the best clinical-pharmacological safety-efficacy profile among the four opioids: oral extended-release morphine, oral extended-release oxycodone, transdermal fentanyl and transdermal buprenorphine. | 15 days after randomization (Reduction of at least 40% of median daily pain, on a NRS)
  We will define a treatment effective if it will produce a mean reduction of NRS values at least of 40% than basal values. Among all effective treatments, we will identify the best as the one that will have a reduction of NRS to a value of 4 or less in 90% of patients compared to the 70% of the others treatments. To evaluate pharmacological safety the plasma concentrations of the drugs and their metabolites will be measured. We will branch patients population in 3 groups to evaluate the correlation between clinical-pharmacological response and genetics (responder,partially and not responder)

SECONDARY OUTCOMES:
Pharmacokinetic of opioids and of their metabolites during long-term administration; correlation between specific genotypes and clinical response or the clinical/pharmacological susceptibility to side-effects on administration of a specific opioid. | 6 months (each patient will be followed for 6 month after enrollment with clinical/pharmacological evaluations once a month and if inefficacy, tolerance or side effects)
  Comparison of plasma levels of opioids and of their metabolites in "responder" patients (clinical effectiveness without side effects), "partially responders" patients (clinical effectiveness without side effects but taking not more than 2 rescue doses per day), and in "non responder" patients (3 groups: clinical un-efficacy, side-effects, tolerance and/or opioid induced hyperalgesia).Evaluation of the correlation between the polymorphisms studied and clinical response; the frequency of allelic variants of interest will be compared in "responder", "partially responder" and "non responder".

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Principal Investigator — IRCCS Foundation Policlinico "San Matteo", Pavia, Italy
Locations (6):
- Italy (6):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - Struttura Complessa di Medicina Interna - Ospedale Civile di Voghera - Azienda Ospedaliera provincia di Pavia, Voghera, Pavia
  - Servizio di Anestesia e Rianimazione e Terapia Antalgica - Ospedale Sant'Orsola-Poliambulanza, Brescia
  - Servizio di Anestesia e Rianimazione e Terapia Antalgica - Ospedale Mellino Mellini, Chiari
  - Unità operativa di Anestesia e Rianimazione - Azienda Ospedaliera San Gerardo, Monza
  - Unità operativa di Terapia Antalgica e Cure Palliative - Ospedale Infermi, Rimini

REFERENCES:
- [Derived] De Gregori S, Minella CE, De Gregori M, Tinelli C, Ranzani GN, Govoni S, Allegri M, Regazzi M. Clinical pharmacokinetics of morphine and its metabolites during morphine dose titration for chronic cancer pain. Ther Drug Monit. 2014 Jun;36(3):335-44. doi: 10.1097/FTD.0000000000000009. PMID 24595069